CLINICAL TRIAL: NCT01299727
Title: An Open-Label Extension of Study HGT-SAN-055 Evaluating Long Term Safety and Clinical Outcomes of Intrathecal Administration of rhHNS in Patients With Sanfilippo Syndrome Type A (MPS IIIA)
Brief Title: Extension of Study HGT-SAN-055 Evaluating Administration of rhHNS in Patients With Sanfilippo Syndrome Type A (MPS IIIA)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Completion of follow-up period
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGT-SAN-067; 2010-021348-16 (EudraCT Number)
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Results first posted 2020-04-21 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: Sanfilippo Syndrome
Keywords: Recombinant Human Heparan N-Sulfatase (rhHNS); Sanfilippo Syndrome Type A (MPS IIIA); Lysosomal storage disease (LSD); Mucopolysaccharidosis (MPS) III
MeSH Terms: conditions — Mucopolysaccharidosis III; Lysosomal Storage Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- rhHNS-10 mg (Experimental): Once per month via an Intrathecal Drug Delivery Device (IDDD) for a maximum of 8 years
  Interventions: Biological: rhHNS-10 mg
- rhHNS-45 mg (Experimental): Once per month via an Intrathecal Drug Delivery Device (IDDD) for a maximum of 8 years
  Interventions: Biological: rhHNS-45 mg
- rhHNS-90 mg (Experimental): Once per month via an Intrathecal Drug Delivery Device (IDDD) for a maximum of 8 years
  Interventions: Biological: rhHNS-90 mg

INTERVENTIONS:
Biological: rhHNS-10 mg — Once per month via an Intrathecal Drug Delivery Device (IDDD) for a maximum of 8 years
  Other Names: Recombinant human heparan N-sulfatase
  Arms: rhHNS-10 mg
Biological: rhHNS-45 mg — Once per month via an Intrathecal Drug Delivery Device (IDDD) for a maximum of 8 years
  Other Names: Recombinant human heparan N-sulfatase
  Arms: rhHNS-45 mg
Biological: rhHNS-90 mg — Once per month via an Intrathecal Drug Delivery Device (IDDD) for a maximum of 8 years
  Other Names: Recombinant human heparan N-sulfatase
  Arms: rhHNS-90 mg

SUMMARY:
Sanfilippo syndrome, or Mucopolysaccharidosis (MPS) III, is a rare lysosomal storage disease (LSD) caused by loss in activity of 1 of 9 enzymes necessary for degradation of the glycosaminoglycan (GAG) heparan sulfate (HS) in lysosomes. MPS IIIA results from deficiency of the enzyme heparan N-sulfatase (sulfamidase). In the absence of this enzyme, intermediates of the HS degradation process accumulate in the lysosomes of neurons and glial cells, with lesser accumulation outside the brain. MPS IIIA symptoms arise on average at 7 months of age, with the average age of diagnosis at 4.5 years for the majority of patients. Patients present a wide spectrum and severity of clinical symptoms. The central nervous system (CNS) is the most severely affected organ system in patients with MPS IIIA, evidenced by deficits in language development, motor skills, and intellectual development. In addition, there are abnormal behaviors including but not limited to aggression and excess motor activity/hyperactivity that contribute to disturbances in sleep.Overall, individuals with MPS IIIA have a marked developmental delay and significantly reduced lifespan to 15 years of age on average.

The purpose of this study is to collect long term safety and tolerability data in patients with MPS IIIA who previously received rhHNS in study HGT-SAN-055 (NCT01155778).

DETAILED DESCRIPTION:
No effective, disease-modifying therapies are currently approved as treatments for this devastating and disabling disease.

Shire Human Genetic Therapies (Shire HGT) is developing a sulfamidase enzyme replacement therapy (ERT)rhHNS for patients with MPS IIIA. rhHNS is being administered into the cerebrospinal fluid (CSF) via an surgically implanted intrathecal drug delivery device (IDDD), because when administered intravenously (IV) it does not cross the blood brain barrier (BBB).

This is a multicenter study designed to collect long-term safety and tolerability data in patients with Sanfilippo Syndrome Type A (MPS IIIA) who received rhHNS via a surgically implanted intrathecal drug delivery device (IDDD) in study HGT-SAN-055 and elected to continue therapy.Patients will continue in the treatment group as they participated in the HGT-SAN-055 study (rhHNS administered by IT injection 10 mg once per month, 45 mg once per month or 90 mg once per month.

The study duration will be a maximum duration of 8 years of rhHNS treatment or until rhHNS is commercially available, the patient discontinues from the study, the Sponsor stops the study, or the Sponsor discontinues the development of rhHNS.

ELIGIBILITY:
Inclusion Criteria:Patients must meet all of the following criteria to be considered eligible for enrollment:

1. The patient must have completed Study HGT SAN 055 and the opinion of the investigator, has no safety or medical issues that contraindicate participation.
2. The patient, patient's parent(s), or legally authorized representative(s) has voluntarily signed an Institutional Review Board / Independent Ethics Committee-approved informed consent form after all relevant aspects of the study have been explained and discussed with the patient's, the patient's, patient's parents or legally authorized representative's consent and patient's assent, as appropriate, must be obtained prior to any study specific procedures.
3. The patient has received at least 5 of the 6 planned infusions of rhHNS in the HGT-SAN-055 study.
4. Patients must be medically stable, in the opinion of the Investigator, to accommodate the protocol requirements, including travel, assessments, and IDDD surgery (if necessary for replacement purposes), without placing an undue burden on the patient/patient's family.

Exclusion Criteria:

Subjects will be excluded from the study if there is evidence of any of the following criteria at screening or at anytime during the study:

1. The patient has experienced an adverse reaction to study drug in Study HGT-SAN-55 that contraindicates further treatment with rhHNS.
2. The patient has a known hypersensitivity to the active ingredient or any excipients in rhHNS drug product.
3. The patient has significant non-MPS IIIA related central nervous system (CNS) impairment or behavioral disturbances that would confound the scientific integrity or interpretation of study assessments, as determined by the Investigator.
4. The patient has significant MPS IIIA behavioral-related issues, as determined by the Investigator, which would preclude performance of study neurocognitive and developmental testing procedures.
5. The patient is pregnant, breast feeding, or is a female patient of childbearing potential, who will not or cannot comply with the use of an acceptable method of birth control, such as condoms, barrier method, oral contraception, etc.
6. The patient has any known or suspected hypersensitivity to anesthesia or is thought to have an unacceptably high risk for anesthesia due to airway compromise or other conditions.
7. The patient has a history of poorly controlled seizure disorder.
8. The patient is currently receiving psychotropic or other medications, which in the Investigator's opinion, would be likely to substantially confound test results and the dose and regimen of which cannot be kept constant throughout the study.
9. The patient cannot sustain absence from aspirin, non-steroidal medications, or medications that affect blood clotting within 1 week prior to a relevant study-related procedure (eg, device re-implantation if applicable), or has ingested such medications within 1 week before any procedures in which any change in clotting activity would be deleterious.
10. The patient has received treatment with any investigational drug (other than rhHNS) intended as a treatment for MPS IIIA within the 30 days prior to, or during the study, or is currently enrolled in another study that involves an investigational drug or device (screening through safety follow-up contact).
11. The patient has received a hematopoietic stem cell or bone marrow transplant.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- Emma Children's Hospital, Academic Medical Center, Amsterdam, Netherlands
- St. Mary's Hospital, Manchester, United Kingdom

REFERENCES:
- [Derived] Wijburg FA, Heap F, Rust S, de Ruijter J, Tump E, Marchal JP, Nestrasil I, Shapiro E, Jones SA, Alexanderian D. Long-term safety and clinical outcomes of intrathecal heparan-N-sulfatase in patients with Sanfilippo syndrome type A. Mol Genet Metab. 2021 Dec;134(4):317-322. doi: 10.1016/j.ymgme.2021.09.003. Epub 2021 Sep 14. PMID 34600820
- [Derived] King B, Marshall N, Beard H, Hassiotis S, Trim PJ, Snel MF, Rozaklis T, Jolly RD, Hopwood JJ, Hemsley KM. Evaluation of enzyme dose and dose-frequency in ameliorating substrate accumulation in MPS IIIA Huntaway dog brain. J Inherit Metab Dis. 2015 Mar;38(2):341-50. doi: 10.1007/s10545-014-9790-8. Epub 2014 Nov 25. PMID 25421091
- [Derived] Langford-Smith A, Wilkinson FL, Langford-Smith KJ, Holley RJ, Sergijenko A, Howe SJ, Bennett WR, Jones SA, Wraith J, Merry CL, Wynn RF, Bigger BW. Hematopoietic stem cell and gene therapy corrects primary neuropathology and behavior in mucopolysaccharidosis IIIA mice. Mol Ther. 2012 Aug;20(8):1610-21. doi: 10.1038/mt.2012.82. Epub 2012 May 1. PMID 22547151

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 2 study centers in the Netherlands and United Kingdom between 01 March 2011 (first participant first visit) and 12 April 2019 (last participant last visit).
Pre-assignment Details: A total of 12 participants were enrolled in this extension study (HGT-SAN-067 [NCT01299727]), with 4 participants included in each of the 3 dose groups. Out of them, 10 participants completed the treatment period of the study.
Groups:
- HGT-1410/rhHNS 10 mg: Participants received HGT-1410/Recombinant human heparan N-sulfatase (rhHNS) 10 milligram (mg) for every 4 weeks (Q4W) via an intrathecal drug delivery device (IDDD).
- HGT-1410/rhHNS 45 mg: Participants received HGT-1410/rhHNS 45 mg for Q4W via IDDD.
- HGT-1410/rhHNS 90 mg: Participants received HGT-1410/rhHNS 90 mg for Q4W via IDDD.
Period: Overall Study
Arm/Group | HGT-1410/rhHNS 10 mg | HGT-1410/rhHNS 45 mg | HGT-1410/rhHNS 90 mg
Started | 4 | 4 | 4
Completed | 0 | 0 | 0
Not Completed | 4 | 4 | 4
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Completed the Treatment Period | 3 | 4 | 3

BASELINE CHARACTERISTICS:
Population: Safety population consisted of all eligible participants from Study HGT-SAN-055 (NCT01155778) who agreed to participate in this extension study, HGT-SAN-067 (NCT01299727). Baseline visit for this study was the first day the participant received their first dose of HGT-1410 in Study HGT-SAN-055 (NCT01155778).
Groups:
- Total: Total of all reporting groups
Arm/Group | HGT-1410/rhHNS 10 mg | HGT-1410/rhHNS 45 mg | HGT-1410/rhHNS 90 mg | Total
Number analyzed (Participants) | 4 | 4 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.145 (4.6956) | 9.070 (9.7916) | 10.638 (8.6645) | 9.618 (7.2941)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 4
  Male | 3 | 2 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 4 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 3 | 3 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) And Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any noxious, pathologic, or unintended change in anatomical, physiologic, or metabolic function as indicated by physical signs, symptoms, or laboratory changes occurring in any phase of a clinical study, whether or not considered study drug related. Treatment-emergent Adverse events (TEAEs) were defined as all adverse events (AEs) from the time of the surgery for first IDDD implantation or first dose of HGT-1410 in study HGT-SAN-055 (NCT01155778) to the data cutoff date, or 30 days after the date of the last dose or 2 weeks after the date of device explant if early termination occurred. TEAEs included participants with any AE, any drug-related AE, any surgery-related AE, any IDDD-related AE, and any IT administration process-related AE, any SAE, any serious drug-related AE.
Time Frame: From start of study drug administration up to follow-up (Month 103)
Population: Safety population consisted of all eligible participants from Study HGT-SAN-055 (NCT01155778) who agreed to participate in this extension study, HGT-SAN-067 (NCT01299727).
Measure: Count of Participants; unit: Participants
Arm/Group | HGT-1410/rhHNS 10 mg | HGT-1410/rhHNS 45 mg | HGT-1410/rhHNS 90 mg
Number analyzed (Participants) | 4 | 4 | 4
Participants
  Participants with at least one TEAEs | 4 | 4 | 4
  Partcipants with at least 1 HGT-1410 Related TEAEs | 4 | 4 | 2
  Participants with at least 1 Surgery Related TEAEs | 4 | 4 | 3
  Participants with at least 1 IDDD Related TEAEs | 4 | 4 | 4
  Participants with at least IT Related TEAEs | 3 | 3 | 2
  Participants with at least 1 Serious TEAEs | 4 | 4 | 3
  Participants with Drug Related Serious TEAEs | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Based on Severity
Description: An adverse event (AE) was any noxious, pathologic, or unintended change in anatomical, physiologic, or metabolic function as indicated by physical signs, symptoms, or laboratory changes occurring in any phase of a clinical study, whether or not considered study drug related. TEAEs were defined as all AEs from the time of the surgery for first IDDD implantation or first dose of HGT-1410 in study HGT-SAN-055 (NCT01155778) to the data cutoff date, or 30 days after the date of the last dose or 2 weeks after the date of device explant if early termination occurred. Severity of an AE is determined by following definitions: Mild: No limitation of usual activities; Moderate: Some limitation of usual activities; Severe: Inability to carry out usual activities.
Time Frame: From start of study drug administration up to follow-up (Month 103)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HGT-1410/rhHNS 10 mg | HGT-1410/rhHNS 45 mg | HGT-1410/rhHNS 90 mg
Number analyzed (Participants) | 4 | 4 | 4
Participants
  Participants with Mild TEAEs | 4 | 4 | 4
  Participants with Moderate TEAEs | 4 | 4 | 3
  Participants with Severe TEAEs | 1 | 2 | 2

3. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities Reported as Treatment Emergent Adverse Events (TEAEs)
Description: Clinical laboratory assessments include hematology, serum chemistry including liver function tests, coagulation urinalysis and cerebrospinal fluid (CSF) were reported.
Time Frame: From start of study drug administration up to follow-up (Month 103)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HGT-1410/rhHNS 10 mg | HGT-1410/rhHNS 45 mg | HGT-1410/rhHNS 90 mg
Number analyzed (Participants) | 4 | 4 | 4
Participants
  Hematology | 2 | 0 | 1
  Serum Chemistry | 1 | 4 | 1
  Urinalysis | 0 | 1 | 1
  Cerebrospinal fluid (CSF) | 3 | 4 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Change in Electrocardiogram (ECG) Reported as Treatment Emergent Adverse Events (TEAEs)
Description: Any change in ECG assessments which were deemed to be clinically significant findings and abnormalities were recorded as TEAEs.
Time Frame: From start of study drug administration up to follow-up (Month 103)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HGT-1410/rhHNS 10 mg | HGT-1410/rhHNS 45 mg | HGT-1410/rhHNS 90 mg
Number analyzed (Participants) | 4 | 4 | 4
Participants | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Postive Anti-rhHNS Antibody Status in Serum by Recombinant Human Heparan N-Sulfatase (rhHNS)
Description: Antibody titers were determined for the samples that tested positive for anti-rhHNS antibodies. Participants with positive Anti-rhHNS antibody status in serum were reported.
Time Frame: Month 103
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HGT-1410/rhHNS 10 mg | HGT-1410/rhHNS 45 mg | HGT-1410/rhHNS 90 mg
Number analyzed (Participants) | 4 | 4 | 4
Participants | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Positive Anti-rhHNS Antibody Status in Cerebrospinal Fluid (CSF) by Recombinant Human Heparan N-Sulfatase (rhHNS)
Description: Antibody titers were determined for the samples that tested positive for anti-rhHNS antibodies. Participants with positive anti-rhHNS antibody in CSF were reported
Time Frame: Month 103
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HGT-1410/rhHNS 10 mg | HGT-1410/rhHNS 45 mg | HGT-1410/rhHNS 90 mg
Number analyzed (Participants) | 4 | 4 | 4
Participants | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline in Bayley Scales of Infant Development Third Edition (BSID-III) at Month 103
Description: BSID-III was used to assess the motor (fine and gross), language (receptive and expressive), and cognitive development of infants and toddlers aged 0-42 months and consisted of a series of developmental play tasks. Score ranges: Cognitive scale 0-91, Receptive communication 0-49, Expressive communication 0-48, Fine motor 0-66 and Gross motor 0-72. Higher values denote stronger skills and abilities in the domain, indicating better outcomes.
Time Frame: Baseline, Month 103
Population: Safety population consisted of all eligible participants from Study HGT-SAN-055 (NCT01155778) who agreed to participate in this extension study, HGT-SAN-067 (NCT01299727). Here, number of participants analyzed signifies participants who were evaluable for this outcome measure at the specific categories.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | HGT-1410/rhHNS 10 mg | HGT-1410/rhHNS 45 mg | HGT-1410/rhHNS 90 mg
Number analyzed (Participants) | 1 | 3 | 2
Score on a scale
  Cognitive: Baseline | 19.00 (NA) — Here, 'NA' indicates that the standard deviation was not calculated as only one participant was evaluated. | 23.33 (12.097) | 21.50 (0.707)
  Cognitive: Change at Month 103: number analyzed (Participants) | 0 | 0 | 1
  Cognitive: Change at Month 103 |  |  | 3.0 (NA) — Here, 'NA' indicates that the standard deviation was not calculated as only one participant was evaluated.
  Receptive: Baseline | 17.00 (NA) — Here, 'NA' indicates that the standard deviation was not calculated as only one participant was evaluated. | 24.00 (16.093) | 17.50 (2.121)
  Receptive: Change at Month 103: number analyzed (Participants) | 0 | 0 | 1
  Receptive: Change at Month 103 |  |  | 0.00 (NA) — Here, 'NA' indicates that the standard deviation was not calculated as only one participant was evaluated.
  Expressive: Baseline | 22.00 (NA) — Here, 'NA' indicates that the standard deviation was not calculated as only one participant was evaluated. | 26.00 (13.528) | 22.50 (0.707)
  Expressive: Change at Month 103: number analyzed (Participants) | 0 | 0 | 1
  Expressive: Change at Month 103 |  |  | 0.00 (NA) — Here, 'NA' indicates that the standard deviation was not calculated as only one participant was evaluated.
  Fine Motor: Baseline | 25.00 (NA) — Here, 'NA' indicates that the standard deviation was not calculated as only one participant was evaluated. | 27.67 (12.423) | 23.50 (2.121)
  Fine Motor: Change at Month 103: number analyzed (Participants) | 0 | 0 | 1
  Fine Motor: Change at Month 103 |  |  | 0.00 (NA) — Here, 'NA' indicates that the standard deviation was not calculated as only one participant was evaluated.
  Gross Motor: Baseline | 21.00 (NA) — Here, 'NA' indicates that the standard deviation was not calculated as only one participant was evaluated. | 26.67 (13.868) | 35.50 (9.192)
  Gross Motor: Change at Month 103: number analyzed (Participants) | 0 | 0 | 1
  Gross Motor: Change at Month 103 |  |  | -21.00 (NA) — Here, 'NA' indicates that the standard deviation was not calculated as only one participant was evaluated.

8. Secondary Outcome: Change From Baseline in Bayley Scales of Infant Development Third Edition (BSID-III)/Kaufman Assessment Battery for Children Second Edition (KABC-II) Age-Equivalent Scores at Month 103
Description: BSID-III was used to assess the motor (fine and gross), language (receptive and expressive), and cognitive development of infants and toddlers aged 0-42 months and consisted of a series of developmental play tasks. KABC-II was an individually administered measure of the processing and reasoning abilities of children and adolescents between the ages of 3 and 18 years and an alternative to BSID-III. Raw scores were converted to age--equivalent scores to measure ability, skill, and knowledge, expressed as the age at which most individuals reach the same level (age norm; range: 0, unbound ). A positive value indicates improvement. The BSID--III and KABC--II age--equivalent scores were based on the cognitive domain and average non-verbal age-equivalent score, respectively.
Time Frame: Baseline, Month 103
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | HGT-1410/rhHNS 10 mg | HGT-1410/rhHNS 45 mg | HGT-1410/rhHNS 90 mg
Number analyzed (Participants) | 2 | 4 | 4
Score on a scale
  Baseline | 66.00 (66.468) | 35.17 (21.678) | 60.90 (60.210)
  Change at Month 103: number analyzed (Participants) | 0 | 0 | 1
  Change at Month 103 |  |  | 3.00 (NA) — Here, 'NA' indicates that the standard deviation was not calculated as only one participant was evaluated.

9. Secondary Outcome: Change From Baseline in Developmental Quotient (DQ) Using Bayley Scales of Infant Development Third Edition (BSID-III) and Kaufman Assessment Battery for Children Second Edition (KABC-II) at Month 103
Description: BSID-III was used to assess the motor (fine and gross), language (receptive and expressive), and cognitive development of infants and toddlers aged 0-42 months and consisted of a series of developmental play tasks. KABC-II was an individually administered measure of the processing and reasoning abilities of children and adolescents between the ages of 3 and 18 years and an alternative to BSID-III. Raw scores of successfully completed items are converted to scale scores and to composite scores. The mean composite score is 100 and the standard deviation (SD) is 15. The DQ was a means to express a neurodevelopmental/cognitive delay which was computed as a ratio and expressed as a percentage using the age equivalent score divided by the age at testing ([age-equivalent score/chronological age] × 100; range: 0-100). A positive value indicates improvement in health and cognition.
Time Frame: Baseline, Month 103
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | HGT-1410/rhHNS 10 mg | HGT-1410/rhHNS 45 mg | HGT-1410/rhHNS 90 mg
Number analyzed (Participants) | 2 | 4 | 4
Score on a scale
  Baseline | 51.91 (27.292) | 43.24 (23.112) | 51.87 (36.095)
  Change at Month 103: number analyzed (Participants) | 0 | 0 | 1
  Change at Month 103 |  |  | -10.96 (NA) — Here, 'NA' indicates that the standard deviation was not calculated as only one participant was evaluated.

10. Secondary Outcome: Change From Baseline in Vineland Adaptive Behavioral Scales Second Edition (VABS-II) at Month 103
Description: VABS-II measured adaptive behaviors, including the ability to cope with environmental changes, to learn new everyday skills, and to demonstrate independence. It was an instrument that supports the diagnosis of intellectual and developmental disabilities in participants. This test measured 5 key domains: communication, daily living skills, socialization, motor skills, and the adaptive behavior composite (a composite of the other four domains). Scoring is 'Usually' = 2, 'Sometimes'/Partially' = 1 or 'Never' = 0. The standard scores represent a score (mean = 100 and standard deviation of 15) on which higher scores indicate a higher level of cognitive ability. A positive change value indicates improvement in adaptive functioning, communication, daily living skills, socialization and motor skills domains were reported here. The range for individual standard scores is 20-160.
Time Frame: Baseline, Month 103
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | HGT-1410/rhHNS 10 mg | HGT-1410/rhHNS 45 mg | HGT-1410/rhHNS 90 mg
Number analyzed (Participants) | 4 | 4 | 4
Score on a scale
  Adaptive Behavior: Baseline | 63.3 (14.61) | 59.0 (26.96) | 59.5 (29.77)
  Adaptive Behavior:Change at Month 103: number analyzed (Participants) | 1 | 0 | 1
  Adaptive Behavior:Change at Month 103 | -18.0 (NA) — Here, 'NA' indicates that the standard deviation was not calculated as only one participant was evaluated. |  | -20.0 (NA) — Here, 'NA' indicates that the standard deviation was not calculated as only one participant was evaluated.
  Communication: Baseline | 68.3 (19.03) | 57.5 (25.94) | 60.3 (30.86)
  Communication: Change at Month 103: number analyzed (Participants) | 1 | 0 | 1
  Communication: Change at Month 103 | -27.0 (NA) — Here, 'NA' indicates that the standard deviation was not calculated as only one participant was evaluated. |  | -20.0 (NA) — Here, 'NA' indicates that the standard deviation was not calculated as only one participant was evaluated.
  Daily Living: Baseline | 62.5 (15.52) | 62.3 (27.58) | 60.0 (30.00)
  Daily Living: Change at Month 103: number analyzed (Participants) | 1 | 0 | 1
  Daily Living: Change at Month 103 | -19.0 (NA) — Here, 'NA' indicates that the standard deviation was not calculated as only one participant was evaluated. |  | -34.0 (NA) — Here, 'NA' indicates that the standard deviation was not calculated as only one participant was evaluated.
  Socialization: Baseline: number analyzed (Participants) | 4 | 4 | 3
  Socialization: Baseline | 64.3 (12.50) | 65.5 (32.42) | 58.7 (35.92)
  Socialization: Change at Month 103: number analyzed (Participants) | 1 | 0 | 0
  Socialization: Change at Month 103 | -15.0 (NA) — Here, 'NA' indicates that the standard deviation was not calculated as only one participant was evaluated. |  |
  Motor Skills: Baseline: number analyzed (Participants) | 3 | 3 | 2
  Motor Skills: Baseline | 82.7 (29.77) | 76.3 (5.69) | 72.5 (12.02)
  Motor Skills: Change at Month 103: number analyzed (Participants) | 1 | 0 | 1
  Motor Skills: Change at Month 103 | -18.0 (NA) — Here, 'NA' indicates that the standard deviation was not calculated as only one participant was evaluated. |  | -14.0 (NA) — Here, 'NA' indicates that the standard deviation was not calculated as only one participant was evaluated.

11. Secondary Outcome: Change From Baseline in Cerebrospinal Fluid (CSF) Total Heparan Sulfate Levels at Month 103
Description: Change from baseline in CSF total heparan sulfate at month 103 was recorded.
Time Frame: Baseline, Month 103
Population: Safety population consisted of all eligible participants from Study HGT-SAN-055 (NCT01155778) who agreed to participate in this extension study, HGT-SAN-067 (NCT01299727). Here, the number of participants analyzed refer to the participants evaluable for this outcome measure at the specific categories.
Measure: Mean (Standard Deviation); unit: micromoles (μmol)
Arm/Group | HGT-1410/rhHNS 10 mg | HGT-1410/rhHNS 45 mg | HGT-1410/rhHNS 90 mg
Number analyzed (Participants) | 4 | 4 | 4
micromoles (μmol)
  Baseline | 5.775 (3.465) | 4.710 (2.968) | 3.795 (1.611)
  Change at Month 103: number analyzed (Participants) | 1 | 0 | 0
  Change at Month 103 | -4.010 (NA) — Here, 'NA' indicates that the standard deviation was not calculated as only one participant was evaluated. |  |

12. Secondary Outcome: Change From Baseline in Urine Glycosaminoglycan (GAG) Levels at Month 103
Description: Change from baseline in Urine GAG at month 103 was recorded.
Time Frame: Baseline, Month 103
Population: Safety population consisted of all eligible participants from Study HGT-SAN-055 (NCT01155778) who agreed to participate in this extension study. Data was not collected for this outcome as the trial was early terminated due to pre-specified efficacy criteria were not met.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | HGT-1410/rhHNS 10 mg | HGT-1410/rhHNS 45 mg | HGT-1410/rhHNS 90 mg
Number analyzed (Participants) | 4 | 4 | 4
microgram per milliliter (mcg/mL) | NA (NA) — Here, 'NA' indicates that the data was not collected due to early termination of the study. | NA (NA) — Here, 'NA' indicates that the data was not collected due to early termination of the study. | NA (NA) — Here, 'NA' indicates that the data was not collected due to early termination of the study.

13. Secondary Outcome: Change From Baseline in Brain Magnetic Resonance Imaging (MRI) at Month 103
Description: Brain MRI parameters include grey matter volume (GMV), white matter volume (WMV) and Intracranial cerebrospinal fluid Volume (ICSFV). Change from baseline in brain MRI at Month 103 was reported.
Time Frame: Baseline, Month 103
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Arm/Group | HGT-1410/rhHNS 10 mg | HGT-1410/rhHNS 45 mg | HGT-1410/rhHNS 90 mg
Number analyzed (Participants) | 4 | 4 | 4
milliliter (mL)
  GMV: Baseline | 550.50 (111.043) | 534.25 (117.291) | 600.28 (67.884)
  GMV: Change at Month 103: number analyzed (Participants) | 1 | 0 | 0
  GMV: Change at Month 103 | -99.49 (NA) — Here, 'NA' indicates that the standard deviation was not calculated as only one participant was evaluated. |  |
  WMV: Baseline | 403.72 (105.575) | 348.28 (76.854) | 442.45 (79.814)
  WMV: Change at Month 103: number analyzed (Participants) | 1 | 0 | 0
  WMV: Change at Month 103 | -33.19 (NA) — Here, 'NA' indicates that the standard deviation was not calculated as only one participant was evaluated. |  |
  ICSFV: Baseline | 26.152 (9.2975) | 22.904 (20.8459) | 20.925 (15.9681)
  ICSFV: Change at Month 103: number analyzed (Participants) | 1 | 0 | 0
  ICSFV: Change at Month 103 | 18.753 (NA) — Here, 'NA' indicates that the standard deviation was not calculated as only one participant was evaluated. |  |

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to follow-up (Month 103).
Groups:
- HGT-1410/rhHNS-10 mg: Participants received HGT-1410/Recombinant human heparan N-sulfatase (rhHNS) 10 milligram (mg) for every 4 weeks (Q4W) via an intrathecal drug delivery device (IDDD).
- HGT-1410/rhHNS-45 mg: Participants received HGT-1410/rhHNS 45 mg for Q4W via IDDD.
- HGT-1410/rhHNS-90 mg: Participants received HGT-1410/rhHNS 90 mg for Q4W via IDDD.
Arm/Group | HGT-1410/rhHNS-10 mg | HGT-1410/rhHNS-45 mg | HGT-1410/rhHNS-90 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 3/4
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HGT-1410/rhHNS-10 mg (N=4) | HGT-1410/rhHNS-45 mg (N=4) | HGT-1410/rhHNS-90 mg (N=4)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Auricular pseudocyst (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Device breakage (General disorders) | 1 (1) | 0 (0) | 0 (0)
Device component issue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Device failure (General disorders) | 2 (2) | 4 (6) | 2 (2)
Device leakage (General disorders) | 1 (1) | 0 (0) | 0 (0)
Device material issue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Central nervous system infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Implant site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
CSF white blood cell count increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Intracranial hypotension (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Medical device change (Surgical and medical procedures) | 3 (6) | 3 (5) | 1 (2)
Medical device removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HGT-1410/rhHNS-10 mg (N=4) | HGT-1410/rhHNS-45 mg (N=4) | HGT-1410/rhHNS-90 mg (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acquired claw toe (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (2)
Growing pains (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Toe walking (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Weight bearing difficulty (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (2) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Ear canal erythema (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (3)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Myopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (8) | 2 (2) | 2 (6)
Defaecation urgency (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (10) | 3 (10) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (2)
Regurgitation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (16) | 3 (23) | 3 (3)
Administration site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter site erythema (General disorders) | 0 (0) | 1 (2) | 0 (0)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter site inflammation (General disorders) | 1 (7) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (2) | 0 (0)
Complication of device insertion (General disorders) | 1 (1) | 0 (0) | 0 (0)
Complication of device removal (General disorders) | 0 (0) | 1 (1) | 0 (0)
Device breakage (General disorders) | 1 (1) | 0 (0) | 0 (0)
Device failure (General disorders) | 1 (1) | 1 (3) | 0 (0)
Device leakage (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (4) | 2 (3) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0)
Implant site effusion (General disorders) | 0 (0) | 1 (1) | 0 (0)
Implant site swelling (General disorders) | 2 (4) | 3 (7) | 2 (3)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Irritability (General disorders) | 3 (4) | 0 (0) | 1 (2)
Local swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 2 (17) | 1 (2) | 1 (7)
Medical device complication (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (18) | 3 (31) | 3 (5)
Thalassaemia trait (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 1 (3) | 0 (0) | 1 (5)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 1 (2)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Abscess oral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Candida nappy rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (6) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Central nervous system infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 2 (3) | 2 (12)
Enterobiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 1 (2) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (4) | 0 (0) | 0 (0)
Helminthic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 1 (2) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (2) | 0 (0) | 1 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (7) | 3 (7) | 2 (4)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (4)
Otitis media (Infections and infestations) | 0 (0) | 2 (2) | 2 (3)
Otitis media acute (Infections and infestations) | 1 (3) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (2) | 1 (1) | 1 (2)
Proteus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 4 (6) | 2 (14) | 3 (5)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 1 (1) | 1 (1)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (2)
Viral rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Drug toxicity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (6) | 1 (1) | 2 (3)
Feeding tube complication (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Nail injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Open wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1)
Procedural site reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Body temperature increased (Investigations) | 1 (2) | 2 (5) | 2 (2)
CSF protein increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
CSF white blood cell count increased (Investigations) | 2 (3) | 3 (3) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (2) | 0 (0)
Lymphocyte count increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Mean cell haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Mean cell volume decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Monocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Norovirus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Red blood cells CSF positive (Investigations) | 0 (0) | 1 (3) | 0 (0)
Serum ferritin decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Enuresis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (5) | 1 (4) | 1 (13)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperphagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Akathisia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Bulbar palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (6)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Crying (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Drooling (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0)
Head titubation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (13) | 1 (6) | 1 (91)
Hyperreflexia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Intracranial hypotension (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Motor dysfunction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (12) | 1 (12) | 2 (9)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 2 (3) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Infection prophylaxis (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Medical device removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 2 (2)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 2 (3) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Conversion disorder (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Obsessive-compulsive disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 2 (3) | 1 (2) | 1 (1)
Sleep disorder (Psychiatric disorders) | 2 (6) | 1 (1) | 0 (0)
Stereotypy (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (3) | 0 (0) | 0 (0)
Labia enlarged (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Penile adhesion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Penile erythema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 1 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (10) | 1 (1) | 1 (7)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 2 (5) | 2 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Eczema (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Scar (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin chapped (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Activities of daily living impaired (Social circumstances) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated as pre-specified efficacy criteria were not met. Data was not presented for efficacy parameters: ABR, Children's Sleep Habits Rating Scale, Infant Toddler QoL Questionnaire, SBRS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT01299727/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/27/NCT01299727/SAP_001.pdf